CLINICAL TRIAL: NCT00815971
Title: Mutations in the Epidermal Growth Factor Receptor(EGFR) Gene in Non-Small Cell Lung Carcinoma (NSCLC) and the Relation to Response of Treatment With Erlotinib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); The Ministry of Science, Technology and Innovation, Denmark (Other Government); Hoffmann-La Roche (Industry)
Responsible Party: PhD, MD Peter Meldgaard and MD Britta Weber, Aarhus University Hospital
Other Study IDs: M-20080012 (ethics committee)
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR mutations; EGFR inhibitor; erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a fine neddle biopsi taken when the diagnosis non-small cell lung carcinoma was made + severals blood samples taken before and during treatment with erlotinib.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSCLC: Patients with non-small cell lung cancer carcinoma treated with erlotinib

SUMMARY:
Recently it has been suggested that specific mutations in the EGFR gene in lung cancer patients is associated with response to a novel drug targeting the EGF system. Recent research also indicates that there is a possible association to the degree of aggressiveness of the disease.

The importance of these mutations is controversial, because the data are based on small studies with highly selected patients.

In this project the investigators want to study the types and frequencies of EGFR mutations in both untreated and treated patients in a systematic manner and relate this to survival.

The thorough registration of patient data in DK enables us to create a strong The investigators expect this knowledge to be of greatest importance for future rational use of drugs targeting the EGF receptors.

DETAILED DESCRIPTION:
Aim:

1. To establish a method for identifying the mutations in the EGFR gene in small clinical samples from lung cancer patients.
2. In a retrospective study(n=500) relate survival to the frequency and types of mutations in the EGFR gene in a Danish population of patients with advanced, inoperable non small cell lung cancer (NSCLC) diagnosed prior to the introduction of treatment directed towards EGFR.
3. In a prospective study (n=300), to identify the mutations in the EGFR gene in patients treated with erlotinib, a tyrosine kinase inhibitor targeting the EGFR. Presence of mutations will be related to the expression of other parts of the EGF system, to mutations in the gene coding for K-RAS and to treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are starting treatment with erlotinib and who has who has signed the informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer who will start treatment with erlotinib
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year after the last patient is enrolled

SECONDARY OUTCOMES:
response( according to RECIST) | 3 month after the last patient is enrolled
quality of live ( measured by EORTC PAL 15) | 3 month after the last patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Peter Meldgaard, PhD MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- department of oncology, University Hospital of Aarhus, Nørrebrogade 44, 8000 Aarhus, Denmark

REFERENCES:
- [Derived] Sorensen BS, Wu L, Wei W, Tsai J, Weber B, Nexo E, Meldgaard P. Monitoring of epidermal growth factor receptor tyrosine kinase inhibitor-sensitizing and resistance mutations in the plasma DNA of patients with advanced non-small cell lung cancer during treatment with erlotinib. Cancer. 2014 Dec 15;120(24):3896-901. doi: 10.1002/cncr.28964. Epub 2014 Aug 7. PMID 25103305
- [Derived] Weber B, Meldgaard P, Hager H, Wu L, Wei W, Tsai J, Khalil A, Nexo E, Sorensen BS. Detection of EGFR mutations in plasma and biopsies from non-small cell lung cancer patients by allele-specific PCR assays. BMC Cancer. 2014 Apr 28;14:294. doi: 10.1186/1471-2407-14-294. PMID 24773774